CLINICAL TRIAL: NCT04410913
Title: Pilot Trial of Visual Healing®, a Nature-themed Virtual Immersive Experience, to Optimize Set and Setting in Psilocybin-assisted Therapy for Alcohol Use Disorder
Brief Title: Pilot Trial of Visual Healing® in Psilocybin-assisted Therapy for Alcohol Use Disorder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keith Heinzerling (Other)
Responsible Party: Sponsor-Investigator, Keith Heinzerling, Director, Pacific Treatment & Research In Psychedelics Program, Saint John's Cancer Institute
Organization: Saint John's Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTRIP002
Record Dates: First submitted 2020-05-18; First posted 2020-06-01 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Alcohol Use Disorder
Keywords: Psilocybin; Psychedelics; Alcohol Use Disorder; Alcoholism; Psychedelic-assisted Therapy
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual Healing Set and Setting (Experimental): Participants in this group will receive a single 25 mg dose of open-label psilocybin along with the Visual Healing Set and Setting protocol. Psilocybin is administered orally as a capsule and taken with water. Four weeks later all participants will undergo a second open-label psilocybin 25 mg session where participants will choose to receive Visual Healing or standard Set and Setting procedures. All participants will receive Prep and Integration counseling.
  Interventions: Drug: Psilocybin plus Visual Healing Set and Setting
- Standard Set and Setting (Active Comparator): Participants in this group will receive a single 25 mg dose of open-label psilocybin along with the Standard Set and Setting protocol. Psilocybin is administered orally as a capsule and taken with water. Four weeks later all participants will undergo a second open-label psilocybin 25 mg session where participants will choose to receive Visual Healing or standard Set and Setting procedures. All participants will receive Prep and Integration counseling.
  Interventions: Drug: Psilocybin plus Standard Set and Setting

INTERVENTIONS:
Drug: Psilocybin plus Visual Healing Set and Setting — Psychedelic session (psilocybin 25 mg) with a therapist who will guide and accompany participants before, during, and after the psychedelic session. In addition, participants will have the chance to view nature-themed videos before and after the psychedelic sessions. Four weeks later, a second psychedelic session (psilocybin 25 mg) with either Visual Healing or standard Set and Setting procedures (patient's choice).
  Arms: Visual Healing Set and Setting
Drug: Psilocybin plus Standard Set and Setting — Psychedelic session (psilocybin 25 mg) with a therapist will guide and accompany participants before, during, and after the psychedelic session. Four weeks later, a second psychedelic session (psilocybin 25 mg) with either Visual Healing or standard Set and Setting procedures (patient's choice).
  Arms: Standard Set and Setting

SUMMARY:
Twenty participants, age 18 or older, who meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for moderate to severe Alcohol Use Disorder will be randomized to open-label psilocybin (25 mg) therapy with the Visual Healing Set and Setting platform (N=10) versus psilocybin (25 mg) with a standard Set and Setting platform (N=10). The purpose of this study is to evaluate the feasibility, safety, and tolerability of adding Visual Healing, a nature-themed virtual immersive program, to psilocybin-assisted therapy among participants with alcohol use disorder.

DETAILED DESCRIPTION:
The objective of the study is to test a strategy for optimizing Set and Setting for psilocybin-assisted therapy of alcohol use disorder. Psilocybin shows promise in early trials for alcohol use disorder, but initial results suggest that patients with alcohol use disorder may be less likely to achieve a mystical experience with standard doses of psilocybin. Optimizing Set and Setting for the psilocybin experience may improve outcomes without requiring higher drug doses. The current study will complete a pilot randomized clinical trial to assess the feasibility, safety, and tolerability of Visual Healing Set and Setting (N=10) versus standard Set and Setting procedures (N=10) in participants with alcohol use disorder undergoing open-label psilocybin 25 mg therapy. In the Visual Healing condition, participants will view nature-themed video programs during the Prep session and during the Ascent phase of the psilocybin experience. Anecdotal reports and reviews suggest that viewing Visual Healing creates a tranquil and calming environment that fosters a stronger connection between the viewer and nature. Psilocybin increases the users feeling of connection to nature and having an intention to connect with nature during the psychedelic session is associated with better outcomes of psychedelic-assisted therapy in initial studies. Reducing pre-dosing anxiety/apprehension and enhancing connections to nature with Visual Healing may improve outcomes of psychedelic-assisted therapy without the need for higher psilocybin doses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to read, speak, and understand English
* Alcohol use disorder, moderate-severe, according to DSM-5 criteria
* Interested in stopping or reducing alcohol use
* Able and willing to adhere to study requirements, including attending all study visits, preparatory, and follow-up sessions, and completing all study evaluations
* Able to swallow capsules
* Women of childbearing potential (WOCBP) must agree to practice an effective means of birth control throughout the duration of the study
* Have an identified support person
* Agree to be driven home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing

Exclusion Criteria:

* Alcohol withdrawal requiring medical intervention
* Women who are pregnant, or women who intend to become pregnant during the study or who are currently nursing
* Unwilling or unable to discontinue formal alcohol use disorder treatment
* Significant current or history of cardiovascular condition
* Have a history of stroke or Transient Ischemic Attack (TIA)
* Moderate to severe liver impairment
* Epilepsy
* Insulin-dependent diabetes
* Diabetes and taking oral hypoglycemic agent with a history of hypoglycemia requiring serious medical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment Rate | Week 10
  Enroll at least 70% of target number of participants
Feasibility: Retention Rate | week 10
  Participants complete at least 70% of post-randomization visits
Tolerability: Number of Visual Healing segments viewed by participants | Week 7
  Average number of segments viewed
Safety/Tolerability: number of Adverse Events | Week 14
  Average number of adverse events (side effects)
Safety: Systolic Blood Pressure | Week 14
  Systolic blood pressure during dosing sessions
Safety: Diastolic Blood Pressure | Week 14
  Diastolic blood pressure during dosing sessions
Safety: Heart rate | Week 14
  Heart rate during dosing sessions
Tolerabilty: Spielberger State-Trait Anxiety Inventory -Short Form (STAI-SF) mean score | Week 14
  Average change in anxiety scale score from prep session to dosing session
Safety: Challenging Experience Questionnaire (CEQ) | Week 14
  Average score on challenging psychedelic experience scale
Safety: Questionnaire for Psychotic Experiences | Week 14
  Average score on psychosis symptom scale

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific Treatment & Research in Psychedelics, Santa Monica, California, United States

REFERENCES:
- [Background] Bogenschutz MP, Forcehimes AA, Pommy JA, Wilcox CE, Barbosa PC, Strassman RJ. Psilocybin-assisted treatment for alcohol dependence: a proof-of-concept study. J Psychopharmacol. 2015 Mar;29(3):289-99. doi: 10.1177/0269881114565144. Epub 2015 Jan 13. PMID 25586396
- [Background] Bogenschutz MP, Podrebarac SK, Duane JH, Amegadzie SS, Malone TC, Owens LT, Ross S, Mennenga SE. Clinical Interpretations of Patient Experience in a Trial of Psilocybin-Assisted Psychotherapy for Alcohol Use Disorder. Front Pharmacol. 2018 Feb 20;9:100. doi: 10.3389/fphar.2018.00100. eCollection 2018. PMID 29515439
- [Background] Brown RT, Nicholas CR, Cozzi NV, Gassman MC, Cooper KM, Muller D, Thomas CD, Hetzel SJ, Henriquez KM, Ribaudo AS, Hutson PR. Pharmacokinetics of Escalating Doses of Oral Psilocybin in Healthy Adults. Clin Pharmacokinet. 2017 Dec;56(12):1543-1554. doi: 10.1007/s40262-017-0540-6. PMID 28353056
- [Background] Carbonaro TM, Bradstreet MP, Barrett FS, MacLean KA, Jesse R, Johnson MW, Griffiths RR. Survey study of challenging experiences after ingesting psilocybin mushrooms: Acute and enduring positive and negative consequences. J Psychopharmacol. 2016 Dec;30(12):1268-1278. doi: 10.1177/0269881116662634. Epub 2016 Aug 30. PMID 27578767
- [Background] Carhart-Harris RL, Bolstridge M, Day CMJ, Rucker J, Watts R, Erritzoe DE, Kaelen M, Giribaldi B, Bloomfield M, Pilling S, Rickard JA, Forbes B, Feilding A, Taylor D, Curran HV, Nutt DJ. Psilocybin with psychological support for treatment-resistant depression: six-month follow-up. Psychopharmacology (Berl). 2018 Feb;235(2):399-408. doi: 10.1007/s00213-017-4771-x. Epub 2017 Nov 8. PMID 29119217
- [Background] Dos Santos RG, Bouso JC, Alcazar-Corcoles MA, Hallak JEC. Efficacy, tolerability, and safety of serotonergic psychedelics for the management of mood, anxiety, and substance-use disorders: a systematic review of systematic reviews. Expert Rev Clin Pharmacol. 2018 Sep;11(9):889-902. doi: 10.1080/17512433.2018.1511424. Epub 2018 Aug 23. PMID 30102078
- [Background] Griffiths RR, Johnson MW, Carducci MA, Umbricht A, Richards WA, Richards BD, Cosimano MP, Klinedinst MA. Psilocybin produces substantial and sustained decreases in depression and anxiety in patients with life-threatening cancer: A randomized double-blind trial. J Psychopharmacol. 2016 Dec;30(12):1181-1197. doi: 10.1177/0269881116675513. PMID 27909165
- [Background] Hasler F, Bourquin D, Brenneisen R, Bar T, Vollenweider FX. Determination of psilocin and 4-hydroxyindole-3-acetic acid in plasma by HPLC-ECD and pharmacokinetic profiles of oral and intravenous psilocybin in man. Pharm Acta Helv. 1997 Jun;72(3):175-84. doi: 10.1016/s0031-6865(97)00014-9. PMID 9204776
- [Background] Johnson M, Richards W, Griffiths R. Human hallucinogen research: guidelines for safety. J Psychopharmacol. 2008 Aug;22(6):603-20. doi: 10.1177/0269881108093587. Epub 2008 Jul 1. PMID 18593734
- [Background] Johnson MW, Griffiths RR. Potential Therapeutic Effects of Psilocybin. Neurotherapeutics. 2017 Jul;14(3):734-740. doi: 10.1007/s13311-017-0542-y. PMID 28585222
- [Background] Johnson MW, Griffiths RR, Hendricks PS, Henningfield JE. The abuse potential of medical psilocybin according to the 8 factors of the Controlled Substances Act. Neuropharmacology. 2018 Nov;142:143-166. doi: 10.1016/j.neuropharm.2018.05.012. Epub 2018 Jun 5. PMID 29753748